CLINICAL TRIAL: NCT07009925
Title: Ivonescimab Combined With Polymeric Micelles Paclitaxel(Pm-Pac) and Platinum (Cisplatin/Carboplatin) as First-line Treatment for Patients With Advanced Squamous NSCLC: A Multicenter, Open-label, Single-arm Clinical Study.
Brief Title: Phase II Study of Platinum (Cisplatin/Carboplatin)and Polymeric Micelles Paclitaxel(Pm-Pac) With Ivonescimab in First Line Metastatic Squamous NSCLC.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Meiqi Shi, chief physician, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MShi
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Squamous Cell Lung Cancer
Keywords: Ivonescimab; Polymeric Micelles paclitaxel; metastatic squamous cell lung cancer; Treatment Outcome; safety

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivonescimab 20mg/kg combined with polymeric micelles paclitaxel and platinum in squamous NSCLC (Experimental)
  Interventions: Drug: Ivonescimab 20mg/kg intravenous every 3 weeks

INTERVENTIONS:
Drug: Ivonescimab 20mg/kg intravenous every 3 weeks — Ivonescimab(20mg/kg) combined with paclitaxel polymeric micelles (≤300mg/㎡) and platinum(cisplatin 75mg/㎡or carboplatin AUC5) IV every 3 weeks for 4 cycles.If patient assessment is of clinical benefit, maintenance therapy with ivonescimab or plus polymeric micelles paclitaxel(≤230mg/m^2) can be continued based on investigator's evaluation and patient's own choice until disease progression or unacceptable toxicity. Ivonescimab is administered first, followed by paclitaxel polymeric micelles and platinum.The maximum treatment duration of ivonescimab and polymeric micelles paclitaxel is 24 months.
  Other Names: paclitaxel polymeric micelles ≤300mg/㎡intravenous every 3 weeks; platinum intravenous every 3 weeks

SUMMARY:
This is a prospective, single-arm, multi-center, phase Ⅱ trial to evaluate the efficacy and safety of Polymeric Micelles paclitaxel(pm-Pac), platinum (cisplatin/carboplatin) in combination with Ivonescimab as first-line treatment in metastatic squamous NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be signed before implementing any trial-related procedures;
2. Age ≥18 years old;
3. Patients with histologically or cytologically confirmed metastatic or recurrent (stage IV) squamous NSCLC (International Association for the Study of Lung Cancer and American Joint Committee on Classification of Cancer, 8th Edition TNM staging), inoperable or inappropriate for radical concurrent chemoradiotherapy, and without previous systemic treatment；. Patients with mixed histology (example adenosquamous) are allowed if there is squamous component in the specimen. PD-L1 immunohistochemical results is required before enrollment.

5.According to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1), there is at least one measurable lesion.

6.Have not received any previous systemic antitumor therapy for advanced/metastatic diseases. Participants who have previously received platinum-based adjuvant/neoadjuvant chemotherapy, or radical chemoradiotherapy for advanced disease are allowed to enroll if the interval between disease progression or recurrence and the end of the last chemotherapy treatment is at least 6 months.

7.ECOG score: 0-1 8.Expected survival time > 3 months 9.Normal organ function, patients should meet the following laboratory indicators:

1. Blood routine test should meet the following criteria (no blood transfusion, no use of blood products, granulocyte colony-stimulating factor, or other hematopoietic growth factors within 7 days before blood routine test); White blood cell count ≥3.0x10^9/L, absolute neutrophil count (ANC) ≥1.5x10^9/L，Platelet count ≥100×10^9/L Hemoglobin >9g/dL. If patients receive blood component transfusion (red blood cells, platelets, etc.) during the screening period, blood routine test should be performed again at an interval of 1 week to meet the above criteria before continuing screening.
2. Blood biochemical examination must meet the following criteria: Total bilirubin ≤1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP) ≤2.5 times ULN (ALT, AST, or ALP≤ 5×ULN for patients with liver metastases, and ALP≤10×ULN for patients with bone metastases); Serum creatinine ≤1.5 times ULN and creatinine clearance (calculated using Cockcroft-Gault formula) ≥60 ml/min；
3. Normal coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
4. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. Subjects with baseline TSH beyond the normal range, but total T3 (or FT3) and FT4 are within the normal range can also be enrolled;
5. Myocardial zymogram within the normal range (if the investor judges that the simple laboratory result is not of clinical significance, the patient is allowed to be included); 10.For female patients of childbearing age, a negative urine or serum pregnancy test should be performed within 3 days before the first study drug administration (day 1 of cycle 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is requested. Female patients who are not of childbearing age are defined as those who have been postmenopausal for at least 1 year or have undergone surgical sterilization or hysterectomy; 11.If there is a risk of conception, all patients (male or female) are required to use contraception throughout the treatment period until 180 days after the last study drug administration.

Exclusion Criteria:

1. Currently participating in interventional clinical research treatment;
2. Has non-squamous histology NSCLC. Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the subject is ineligible; for non-small cell histology if there is any squamous element is present (example adenosquamous), the subject is eligible; the squamous element does not have to be predominant.
3. Previously received immunotherapy, including immune checkpoint inhibitors (such as anti-PD-1 /L1 antibodies, anti-CTLA-4 antibodies, anti-LAG-3 antibodies, etc.), immune checkpoint agonists (such as: Subjects of ICOS, CD40, CD137, GITR, OX40 antibody, etc.), immune cell therapy, etc., any treatment targeting the immune mechanism of tumor action;
4. known allergic or hypersensitive reactions to any investigational drug or any excipients thereof;
5. Have a history of severe bleeding or coagulopathy; Clinically significant bleeding symptoms, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing up or spitting up ≥1 TSP of blood or small blood clots or only coughing up blood with no sputum, allowing inclusion of blood in the sputum), nasal bleeding (excluding nosebleed and retractive rhinorrhea) within 1 month before first administration; Imaging during the screening period showed that the tumor surrounded important blood vessels or had obvious necrosis and voids, and the researchers determined that entering the study would cause bleeding risk. Central, squamous non-small cell lung cancer with cavities and a higher risk of bleeding as determined by the investigators; Received continuous antiplatelet or anticoagulant therapy within 10 days prior to initial administration;
6. Tumor invasion of surrounding important organs and blood vessels (such as aorta, heart and pericardium, superior vena cava, trachea, esophagus, etc.) or esophagotracheal fistula or esophagopleural fistula risk;
7. Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (subjects who do not require drainage effusion or whose frequency of drainage is less than once per month can be enrolled);
8. Patients with symptomatic brain metastases, meningeal metastases, or spinal cord compression;
9. There is a history or current presence of non-infectious pneumonia/interstitial lung disease requiring systemic glucocorticoid therapy;
10. Serious comorbidities such as a history of severe lung or heart disease, any arterial thrombosis, embolism, or ischemia within 6 months prior to treatment, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack. A history of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within the 3 months prior to enrollment (implantable intravenous port or catheter-derived thrombosis, or superficial venous thrombosis was not considered "severe" thromboembolism);
11. History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with autoimmune related hypothyroidism receiving stable dose thyroid hormone replacement therapy were eligible to participate in the study. Patients with controlled type 1 diabetes following a stable insulin regimen were eligible to participate in the study.
12. Active systemic infections, including tuberculosis (clinical diagnosis including clinical history, physical examination and imaging findings, and TB testing based on local medical practice), hepatitis B (known to be positive for HBV surface antigen (HBsAg), HBV DNA ≥1000cps/ml or the lower limit of its reference value), hepatitis C or human immunodeficiency virus (HIV antibody positive);
13. A known mental illness or substance abuse condition that may affect compliance with the test requirements;
14. There is a medical history, disease, treatment, or abnormal laboratory result that could interfere with the test results or prevent the subject from fully participating in the study, or the investigator believes that participation in the study is not in the subject's best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | From the start of treatment until disease progression or death (assessed up to 24 months)
  Progression-free Survival (PFS) is defined as the time from the first study dose date to the date of first documentation of disease progression or death (whichever occurred first) based on RECIST 1.1 assessed by investigator review.

SECONDARY OUTCOMES:
Objective Response Rate | Every 6 weeks (RECIST 1.1) until progression (up to 24 months)
  Objective Response Rate (ORR) Based on RECIST 1.1 assessed by investigator review, the proportion (%) of patients with confirmed best overall response of complete response (CR) or partial response (PR).
Disease Control Rate | From the first dose of study drug to the first date of documentation of disease progression or death whichever occurred first, up to approximately 2 years
  Disease Control Rate (DCR) Based on RECIST 1.1 assessed by investigate review ,the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR), or stable disease (SD).
Duration of Response | From date of first documented confirmed CR or PR until date of first documentation of PD or death whichever occurred first, up to approximately 2 years
  Duration of Response (DOR) is defined as the time from the first documentation of CR or PR to the date of first documentation of PD or death (whichever occurred first) in participants with confirmed CR or PR based on RECIST 1.1 assessed by investigator review
Overall Survival | From the date of first dose of study drug until date of death from any cause (up to approximately 5 years )
  Overall Survival (OS) was measured from the date of first dose of study drug until date of death from any cause.Participants who were lost to follow-up and the participants who were alive at the date of data cutoff was censored at the date the participant was last known alive, whichever came earlier
Incidence of Adverse Events | From first dose until 30 days after the last dose, up to approximately 2 years.
  Number of Participants With adverse events (AE), Treatment-releated Adverse Events (TRAEs), Serious Adverse Events (SAEs) and immune-related adverse events (irAE), events will be classified according to CTCAE V5.0.

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to external researchers due to patient privacy constraints, contractual agreements with sponsors.

REFERENCES:
- [Background] Xiong A, Wang L, Chen J, Wu L, Liu B, Yao J, Zhong H, Li J, Cheng Y, Sun Y, Ge H, Yao J, Shi Q, Zhou M, Chen B, Han Z, Wang J, Bu Q, Zhao Y, Chen J, Nie L, Li G, Li X, Yu X, Ji Y, Sun D, Ai X, Chu Q, Lin Y, Hao J, Huang D, Zhou C, Shan J, Yang H, Liu X, Wang J, Shang Y, Mei X, Yang J, Lu D, Hu M, Wang ZM, Li B, Xia M, Zhou C. Ivonescimab versus pembrolizumab for PD-L1-positive non-small cell lung cancer (HARMONi-2): a randomised, double-blind, phase 3 study in China. Lancet. 2025 Mar 8;405(10481):839-849. doi: 10.1016/S0140-6736(24)02722-3. PMID 40057343
- [Background] HARMONi-A Study Investigators; Fang W, Zhao Y, Luo Y, Yang R, Huang Y, He Z, Zhao H, Li M, Li K, Song Q, Du X, Sun Y, Li W, Xu F, Wang Z, Yang K, Fan Y, Liu B, Zhao H, Hu Y, Jia L, Xu S, Yi T, Lv D, Lan H, Li M, Liang W, Wang Y, Yang H, Jia Y, Chen Y, Lu J, Feng J, Liu C, Zhou M, Zhou J, Liu X, Zhou N, He M, Dong X, Chen H, Chen Y, Su H, Li X, Zhang Z, Yang L, Cheng Y, Chen L, Hou X, Zhang Y, Guo J, Wang Z, Lu H, Wu D, Feng W, Li W, Huang J, Wang Y, Song X, Peng J, Liu L, Guo Y, Li W, Lu D, Hu M, Wang ZM, Li B, Xia M, Zhang L. Ivonescimab Plus Chemotherapy in Non-Small Cell Lung Cancer With EGFR Variant: A Randomized Clinical Trial. JAMA. 2024 Aug 20;332(7):561-570. doi: 10.1001/jama.2024.10613. PMID 38820549
- [Background] Socinski MA, Nishio M, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Kong S, Lee A, Coleman S, Zou W, McCleland M, Shankar G, Reck M. IMpower150 Final Overall Survival Analyses for Atezolizumab Plus Bevacizumab and Chemotherapy in First-Line Metastatic Nonsquamous NSCLC. J Thorac Oncol. 2021 Nov;16(11):1909-1924. doi: 10.1016/j.jtho.2021.07.009. Epub 2021 Jul 24. PMID 34311108
- [Background] Boyd JA, Hubbs JL, Kim DW, Hollis D, Marks LB, Kelsey CR. Timing of local and distant failure in resected lung cancer: implications for reported rates of local failure. J Thorac Oncol. 2010 Feb;5(2):211-4. doi: 10.1097/JTO.0b013e3181c20080. PMID 19901853
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Shi M, Gu A, Tu H, Huang C, Wang H, Yu Z, Wang X, Cao L, Shu Y, Wang H, Yang R, Li X, Chang J, Hu Y, Shen P, Hu Y, Guo Z, Tao M, Zhang Y, Liu X, Sun Q, Zhang X, Jiang Z, Zhao J, Chen F, Yu H, Zhang W, Sun J, Li D, Zhou J, Han B, Wu YL. Comparing nanoparticle polymeric micellar paclitaxel and solvent-based paclitaxel as first-line treatment of advanced non-small-cell lung cancer: an open-label, randomized, multicenter, phase III trial. Ann Oncol. 2021 Jan;32(1):85-96. doi: 10.1016/j.annonc.2020.10.479. Epub 2020 Oct 29. PMID 33130217
- [Background] Shi M, Sun J, Zhou J, Yu H, Yu S, Xia G, Wang L, Teng Y, Liu G, Yu C, Feng J, Shen Y. Phase I dose escalation and pharmacokinetic study on the nanoparticle formulation of polymeric micellar paclitaxel for injection in patients with advanced solid malignancies. Invest New Drugs. 2018 Apr;36(2):269-277. doi: 10.1007/s10637-017-0506-4. Epub 2017 Sep 4. PMID 28868573
- [Background] Zhao Y, Chen G, Chen J, Zhuang L, Du Y, Yu Q, Zhuang W, Zhao Y, Zhou M, Zhang W, Zhang Y, Wan Y, Li W, Song W, Wang ZM, Li B, Xia M, Yang Y, Fang W, Huang Y, Zhang L. AK112, a novel PD-1/VEGF bispecific antibody, in combination with chemotherapy in patients with advanced non-small cell lung cancer (NSCLC): an open-label, multicenter, phase II trial. EClinicalMedicine. 2023 Aug 3;62:102106. doi: 10.1016/j.eclinm.2023.102106. eCollection 2023 Aug. PMID 37593227
- [Background] Chen Z, Wu L, Wang Q, Yu Y, Liu X, Ma R, Li T, Li Y, Song X, Li L, Zhao W, Wang Q, Xu X, Lu S. Brief Report: Ivonescimab Combined With Etoposide Plus Carboplatin as First-Line Treatment for Extensive-Stage SCLC: Results of a Phase 1b Clinical Trial. J Thorac Oncol. 2025 Feb;20(2):233-239. doi: 10.1016/j.jtho.2024.10.013. Epub 2024 Oct 28. PMID 39490738
- [Background] Wang L, Luo Y, Ren S, Zhang Z, Xiong A, Su C, Zhou J, Yu X, Hu Y, Zhang X, Dong X, Meng S, Wu F, Hou X, Dai Y, Song W, Li B, Wang ZM, Xia Y, Zhou C. A Phase 1b Study of Ivonescimab, a Programmed Cell Death Protein-1 and Vascular Endothelial Growth Factor Bispecific Antibody, as First- or Second-Line Therapy for Advanced or Metastatic Immunotherapy-Naive NSCLC. J Thorac Oncol. 2024 Mar;19(3):465-475. doi: 10.1016/j.jtho.2023.10.014. Epub 2023 Oct 23. PMID 37879536
- [Background] Frentzas S, Austria Mislang AR, Lemech C, Nagrial A, Underhill C, Wang W, Wang ZM, Li B, Xia Y, Coward JIG. Phase 1a dose escalation study of ivonescimab (AK112/SMT112), an anti-PD-1/VEGF-A bispecific antibody, in patients with advanced solid tumors. J Immunother Cancer. 2024 Apr 19;12(4):e008037. doi: 10.1136/jitc-2023-008037. PMID 38642937
- [Background] Voron T, Colussi O, Marcheteau E, Pernot S, Nizard M, Pointet AL, Latreche S, Bergaya S, Benhamouda N, Tanchot C, Stockmann C, Combe P, Berger A, Zinzindohoue F, Yagita H, Tartour E, Taieb J, Terme M. VEGF-A modulates expression of inhibitory checkpoints on CD8+ T cells in tumors. J Exp Med. 2015 Feb 9;212(2):139-48. doi: 10.1084/jem.20140559. Epub 2015 Jan 19. PMID 25601652